CLINICAL TRIAL: NCT07331389
Title: A Phase I, Single-center, Open-Label, Single-Arm, Fixed-Sequence Study to Evaluate the Drug-Drug Interaction of HDM1002 and Metformin, Empagliflozin, Midazolam, Valsartan, and Warfarin in Overweight/Obese Adult Chinese Subjects
Brief Title: A Drug-Drug Interaction Study of HDM1002 and Metformin, Empagliflozin, Midazolam, Valsartan, and Warfarin
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HDM1002-111
Record Dates: First submitted 2025-11-18; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Overweight Subject; Healthy Subjects
Keywords: HDM1002
MeSH Terms: interventions — Metformin; empagliflozin; Midazolam; Valsartan; Warfarin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- experimental arm (Experimental): Cohort 1 (Study on the Interaction between HDM1002 and Metformin, empagliflozin), Cohort 2 (Study on the Interaction between HDM1002 and Midazolam, valsartan, Warfarin)
  Interventions: Drug: Metformin; Drug: Empagliflozin; Drug: Midazolam; Drug: Valsartan; Drug: Warfarin; Drug: HDM1002

INTERVENTIONS:
Drug: Metformin — Administered orally
Drug: Empagliflozin — Single dose; Administered orally
Drug: Midazolam — Single dose; Administered orally
Drug: Valsartan — Single dose; Administered orally
Drug: Warfarin — Single dose; Administered orally
Drug: HDM1002 — Administered orally

SUMMARY:
The purpose of this study is to characterize the drug-drug intereaction of HDM1002 and metformin, empagliflozin, midazolam, valsartan, and warfarin in overweight/obese adult subjects. The safety and tolerability of HDM1002 with metformin, empagliflozin, midazolam, valsartan, and warfarin when given separately or together will also be evaluated

ELIGIBILITY:
Inclusion Criteria:

1. According to the medical history, clinical laboratory test results, vital sign measurements, 12 lead ECG results, and physical examination results during the screening period, the investigator considers the subject to be in good general health.
2. Age range of 18-45 years old (including range), no limit to gender.
3. Subject weighed ≥50.0 kg, and a body mass index (BMI) within the range of 24.0 - 35.0 kg/m2 (including cut-off values).

Exclusion Criteria:

1. Subject has a history or family history of medullary thyroid cancer, thyroid C-cell hyperplasia, or multiple endocrine neoplasia type 2 (MEN2), or calcitonin≥50 ng/L during the screening period.
2. History of chronic pancreatitis or an episode of acute pancreatitis within 3 months prior to screening.
3. History of acute cholecystitis attack within 3 months prior to screening.
4. Severe hypoglycemic events or recurrent hypoglycemic events occurred within 3 months prior to screening
5. Subject judged by investigator has dysphagia, diseases or conditions that affect gastric emptying, or affect the absorption of gastrointestinal nutrients, such as bariatric surgery or other gastrectomy, irritable bowel syndrome, dyspepsia, etc.
6. Any pre-existing conditions that increase the risk of bleeding, such as acute gastritis or active ulcers with bleeding, hemorrhagic cerebral infarction, epidural hematoma, intracranial hematoma, intraventricular hemorrhage, subarachnoid hemorrhage, and active pathological bleeding, etc
7. History of previous surgery that will affect the absorption, distribution, metabolism, and excretion of drugs or plan to undergo surgery during the study period.
8. During screening period, any abnormalities in physical examination, electrocardiogram, laboratory tests, and vital signs which are of clinically significant .
9. Taken or planned to take any drug that effect liver enzyme or transporter activity within 28 days prior to taking the investigational drug.
10. History of clinically significant cardiovascular and cerebrovascular disease within 6 months prior to screening or at the time of admission.
11. Presence of clinically significant ECG results judged by the investigator at screening.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 111 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2026-01-12 (Estimated); Study Completion 2026-06-13 (Estimated)

PRIMARY OUTCOMES:
AUC[0-∞] | through study completion, an average of 11 weeks
  PK parameter of metformin, empagliflozin, midazolam, valsartan, and warfarin:Area under the curve from time 0 hour to ∞
Cmax | through study completion, an average of 11 weeks
  PK parameter of metformin, empagliflozin, midazolam, valsartan, and warfarin: Maximum observed concentration
AUC[0-t] | through study completion, an average of 11 weeks
  PK parameter of metformin, empagliflozin, midazolam, valsartan, and warfarin: Area under the curve from time 0 to t hour

SECONDARY OUTCOMES:
PK parameter of HDM1002 | through study completion, an average of 11 weeks
  PK parameter of HDM1002 including Tmax, T1/2, CL/F, Vz/F, MRT, etc
other PK parameters | through study completion, an average of 11 weeks
  Other PK parameters of metformin, empagliflozin, midazolam, valsartan, warfarin: Tmax, T1/2, CL/F, Vz/F, MRT, etc
Adverse events (AEs) | through study completion, an average of 11 weeks
  Number of subjects reporting AEs

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Anhui Medical University, Hefei, China